CLINICAL TRIAL: NCT05070377
Title: ActTeens Program: A Program to Improve the Physical Activity Level, Physical Fitness, Cardiometabolic and Mental Health in Adolescents
Brief Title: A Physical Activity Program for Adolescents - ActTeens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antonio Stabelini Neto (Other)
Responsible Party: Sponsor-Investigator, Antonio Stabelini Neto, Professor, Universidade Estadual do Norte do Parana
Organization: Universidade Estadual do Norte do Parana (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ActTeens
Record Dates: First submitted 2021-09-24; First posted 2021-10-07 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: Active Behavior; Muscular Fitness; Cardiorespiratory fitness; Metabolic profile; Well-being; ill-being; Teens
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The ActTeens Program will include interventions in three different context: (1) structured physical activity sessions by physical education (school), (2) self-monitoring plus goal setting by pedometer (out-of-school), and (3) healthy lifestyle guidance (social support). The structured PA will be developed in PE lessons, twice a week, with twenty-minute each lesson (40 min·week) To promote active behavior out-of-school will be used a pedometer plus goals setting where each adolescent of the intervention group will receive their own goal (based on the number of steps measured in the baseline week) outlining the goals to achieve weekly. To improve healthy behavior will be sent by WhatsApp® messages about healthy eating and regular PA for the intervention and parents groups.
  Interventions: Other: Physical activity
- Control (No Intervention): The control group participated in usual practice (regularly scheduled PE and postcurricular school sport) for the duration of the study .

INTERVENTIONS:
Other: Physical activity — 1. structured physical activity sessions by physical education (school), twice a week, with twenty-minute each lesson;
  2. self-monitoring plus goal setting by pedometer (out-of-school), progressive goals to achieve weekly;
  3. healthy lifestyle guidance ( parents social support).
  Arms: Intervention

SUMMARY:
The purpose of this study is to assess the ActTeens (Active teens) Program to improve the physical activity level, physical fitness, cardiometabolic and mental health in adolescents. The investigators hypothesize that that intervention group participant's fitness and physical activity levels will improve during this period in comparison with control group participants.

DETAILED DESCRIPTION:
Introduction The practice of regular physical activity (PA) has been associated with numerous health benefits including improve cardiorespiratory fitness (CRF), body composition, cardiometabolic profile and mental health. Furthermore, evidence suggests that 81% of school-aged adolescents aged 11 to 17 years not meeting the current recommendations, and in Brazil, only 8.4% adolescents are physically active. In Brazil, school-based programs have been developed with a focus on the promotion of active behaviour in teens, however, these programs implemented interventions with strategies only in the school context with predominantly focus on the aerobic component of youth PA guidelines. In addition, a number limit of physical activity programs in the school setting is being conducted in low-and- middle-income countries. Thus, considering PA benefits for health, knowing the need to develop strategies to encourage active behavior both school and out of school, and that few studies of interventions are approach with focusing on muscular fitness (MF). There is a need to implement school-based programs that provide new opportunities for practice in the school setting and promote an active lifestyle outside of school for adolescents.

METHODS Study Design The trial is approved by human research ethics committee of the States University of Northern of Parana (nº 4.452.513). The design, conduct, and reporting will adhere to the guidelines of the Consolidated Standards of Reporting Trials. The intervention will be evaluated using a two-arm school-based randomized clinical trial with one intervention group (IG) and a control group (CG). The assessment will be conducted at baseline, 6 months (primary end).

School recruitment and selection The secondary public schools in Jacarezinho city, including students from 13 - 14 years (i.e., Grade 8 and 9) will be recruited via the list provided by the Regional Education Center of Jacarezinho city, Pr, regarding the 2022 academic year. Then emails will be sent directly to eligible schools (school principals and Grade 8 and 9 coordinators). Each school should provide a list with the number of classes, for Grade 8 and 9, one class of each year education will be randomly selected to participate.

Participants Two grades 8 and 9 (one each year) teachers per school that agree to participate in the program during the scheduled class time, and students.

Sample size calculation The sample size estimation was conducted using G*Power (version 3.1) and based on detecting changes in the primary outcome of physical activity. Based on previous research, the investigators anticipate the effect size for PA of d = 0.25 (an adjusted for baseline of 5 min moderate-to-vigorous physical activity (MVPA) per day and assuming a standard deviation of MVPA of 17.8 minutes with correlation of 0.59 between baseline and follow-up). The researchers adjusted for clustering at the class level using a correction factor of [1 + (m - 1) x ICC], where m represents the number of participants per class and ICC refers to the intraclass correlation coefficient for PA. Assuming an average class size of 29 participating students, two classes per school and an intraclass correlation coefficient (ICC) for PA of 0.034. Allowing for an expected dropout of 20% at the study endpoint, the required sample size to achieve 85% power with alpha levels set at 0.05 is 70 students by schools.

Blinding and Randomisation Randomization will occur among schools that have been recruited and have completed baseline assessments. The schools will be matched based on the following characteristics: school area-level socioeconomic status (i.e., using Socio-Economic Class ABEP). Schools will be randomised to either a control or an intervention condition by independent research using a computer-based random number generator.Afterwards each school will provide a list with the number of classes, one class of each year education (Grade 8 and 9) will be randomly selected to participate. Schools randomised to the intervention condition will the program during the study period, whereas schools allocated to the control condition will continue usual school practice (normal curricular lessons) for the duration of the study period intervention (6-month from baseline). And after the final study assessment, schools allocated to the control group will then receive the intervention.

INTERVENTION The ActTeens Program is a school-based PA intervention, will be developed over one school term (6 months) and will be designed to improve adolescent´s physical activity level, physics, metabolic, and mental health. The ActTeens Program will include interventions in three different context: (1) structured physical activity sessions by physical education (school), (2) self-monitoring plus goal setting by pedometer (out-of-school), and (3) healthy lifestyle guidance (social support). The intervention will be guided by social cognitive theory (SCT) and self-determination theory (SDT) and will target teachers, schools, students and parents.

The structured physical activity(PA) sessions, which focused on resistance training (RT) is an adaptation of the Australian Resistance Training for Teens Program, which originated from Nutrition and Enjoyable Activity for Teen (NEAT) and Active Teen Leaders Avoiding Screen-Time (ATLAS) interventions, and will be designed to satisfy participants' basic psychological needs for autonomy, competence, and relatedness, to support autonomous motivation and self-efficacy for physical activity. The structured PA will be developed in physical education (PE) lessons, twice a week, with twenty-minute each lesson (40 min·week). The implementation strategies used to support adoption and delivery will include: (i) professional learning workshop for teachers; (ii) provision of teacher handbook, session resources and fitness equipment; and (iii) physical activity session observation and feedback. The intervention will consist of the following components: (i) introductory seminar for students delivered by teachers; (ii) a structured physical activity program, which focused on RT by circuit cards (physical education).

The structured physical activity of resistance training will follow specific session format, including: movement-based games and dynamic stretching warm-up; RT skill development; high intensity RT (HIRT) workout. Participants will be able to select from a variety of predesigned RT circuit cards, which will be released across the program to promote variety and sustain participant interest. The level of intensity for each session component will be guided by Borg´s rating of perceived exertion scale.

To promote exercise adherence, physical activity sessions will be developed with a focus on enhancing students' autonomous motivation for RT within and beyond the school setting by satisfying their basic psychological needs for autonomy (feeling in control), competence (feeling capable) and relatedness (feeling connected with others) founded upon the tenets of SDT. Teachers will learn to facilitate RT sessions using the Supportive, Active, Autonomous, Fair, and Enjoyable (SAAFE) teaching principles, which will serve as a framework for design and delivery of the physical activity sessions, as well as observations sessions. Teachers will be educated about the importance of, and provide with strategies of, integrating SAAFE principles in their lessons by learning workshop.

Participants' need for autonomy will be satisfied by providing opportunities for choice within sessions (e.g., type of activity and preferred music playing) and explaining the rationale for the program in an information seminar. The introductory seminar will reinforce the importance of exercise for physical health (focus in muscular fitness), metabolic profile and behavioral change such as physical activity self-monitoring and goal setting. Competence will be satisfied using positive and specific feedback from teachers to enhance self-efficacy (e.g., providing encouragement, giving specific feedback on technique, modelling correct performance). Teachers will be encouraged to adopt practices that support relatedness and group cohesion during RT sessions (i.e., encouraging supportive behaviour among students). Several precautions will be undertaken to ensure the safety of participants including: 1) explanation of correct technique for all exercises in the introductory student seminar session; 2) inclusion of warm-ups and cool-downs; and 3) reminders for teachers and research staff member to monitor and correct exercise technique.

Regarding the sessions, a range of sociocultural targeting strategies will be applied to the interventions to increase their relevance and appeal to adolescent boys and girls. For example, the circuit cards and interactive seminar will include images of females and males-sex role models. In addition, the content of the interactive seminar will be designed to be relevant to boys and girls by recognising and focusing on health behaviors common to each sex. However, the sessions will be conducted with mixed-sex groups.

To promote active behavior out-of-school will be used a pedometer plus goals setting where each adolescent of the intervention group will receive their own goal (based on the number of steps measured in the baseline week) outlining the goals to achieve weekly. The goals will be predetermined by the researcher of way progressive, and also will be sent by WhatsApp® messages to encourage adolescents to practice daily PA. To improve healthy behavior will be sent by WhatsApp® messages about healthy eating and regular PA for the intervention and parents groups. The control group participated in usual practice (regularly scheduled PE and postcurricular school sport)..

Measures and data collection All assessments will be conducted at the study school by trained research assistants, who will be blinded to group allocation at all time-points. Socioeconomic (SES) information and self-report measures using questionnaires and will occur prior to fitness assessment. Anthropometric assessments will be conducted in a sensitive manner by same-sex researcher staff when possible. The research assistants will provide a brief verbal description and demonstration of each fitness test prior to commencement.

STATISTICAL ANALYSES Linear mixed models will be used to analyse the primary and secondary outcomes using Statistical Package for the Social Sciences(SPSS) for Windows (version 20.0; 2010 SPSS Inc, IBM Company, Armonk, NY 2010 SPSS Inc., IBM Company, Armonk, NY), with significance set at P< 0.05. The models will be used to assess the effect of treatment ( IG or control), time (baseline and 24 weeks) and the group-by-time interaction, weighted for sex and adjusted for the covariates maturation and BMI. Mixed model analyses are consistent with the intention-to-treat principle, assuming the data are missing at random. Effect sizes between groups will be calculated using Cohen's d (the adjusted difference between the control and intervention groups over time divided by the pooled standard deviation of change) and interpreted as follows: d = 0.2 (small), d = 0.5 (medium), and d = 0.8(large). Potential moderators will be explored using linear mixed models with interaction terms for the following: sex (male, female), socioeconomic status (low, medium, high), initial weight status (healthy weight vs overweight/obese). Subgroup analyses will be only conducted if significant interaction effects P≤0.10. Hypothesized mediators of physical activity behaviour change will be examined using multilevel linear analysis.

ELIGIBILITY:
Inclusion Criteria:

* Schools: secondary public schools in Jacarezinho city, including students from 13 - 14 years (i.e., Grade 8 and 9); physical education lessons on alternate days.
* Teacher: Two grades 8 and 9 (one each year) teachers per school that agree to participate in the program during the scheduled class time;
* Eligible Adolescents are grade 8 or 9 students with age between 13-14 years whose the parents or legal guardians accept and sign the informed consent authorization the use of their data.

Exclusion Criteria:

* Students with the cardiometabolic disease diagnosed (type 2 diabetes; hypertension) and with a physical or mental condition that would preclude their participation in physical activity program will be excluded from the study (analysis), but will still participate in normal lessons.

Ages: 13 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in physical activity at week 24 | Baseline and week 24
  Adolescents will be instructed to wear an Actigraph (GT3X) accelerometer on the hip at the height of the anterior iliac spine for all day (except when bathing, swimming, sleeping) for a period of seven consecutive days. The subjects who use at least wear time of >8 h on 3 days or more (including 1 weekend) will be included in the valid analyses data. The time (minutes/day) spent in physical activity of different light, moderate and vigorous intensities will be estimated, using validated cut off points. Non-wear time, defined as ≥60 min of continuous '0' counts, will be removed from the dataset. Weekday and weekend days physical activity will be calculated separately (i.e., mean minutes per day).

SECONDARY OUTCOMES:
Change from baseline in cardiometabolic health at week 24 | Baseline and week 24
  The cardiometabolic variables that will be analysed are glucose(mg/dL), triglyceride-TG (mg/dL), total cholesterol-TC (mg/dL) and glycated hemoglobin -HbA1c (mg/dL) by blood samples.
Change from baseline in insulin at week 24 | Baseline and week 24
  The cardiometabolic variable that will be analysed is insulin ((μUI/mL) by blood samples.
Change from baseline in muscular fitness at week 24 | Baseline and week 24
  Upper body muscular and lower body muscular endurance will be assessed using a 90-degree push-up(reps) and sit-to-stand test (reps), respectively. In the 90-degree push-up test, the participant should do push-up until a 90-degree angle is formed at the elbow before pushing back up, using a cadence of 40 beats per minute. The test will be concluded when the participant either fails to do a push-up in the angle required on two non-consecutive repetitions (warning verbalised by an assessor, repetitions counted), fails to maintain movement in time with the metronome, fails to maintain appropriate technique (back straight) or on the volitional failure of the test. To lower body muscular endurance, the volunteer will sit in a chair (regardless of the height of the participant) with his back against the back of the chair. The students will be asked to go from a sitting to a standing position and back to a sitting position for 30 seconds as many times as possible.
Change from baseline in cardiorespiratory fitness at week 24 | Baseline and week 24
  CRF will be assessed using PACER FITNESSGRAM test and will be administered following standardized procedures, which have excellent validity and reliability in this population. Test administrators will provide verbal encouragement during the shuttle to maximise participant motivation. A 20m course will be set up on a hard surface with participants instructed to run back and forth between two sets of lines while keeping pace with a pre-recorded cadence (indicated by a single beep for each 20m shuttle). The test will be terminated when the participants fail to complete two consecutive laps in the allotted time or voluntarily dropped out due to fatigue.
Change from baseline in anxiety, depression and stress symptoms on the Depression and Anxiety Stress Scale-short form (DASS 21) at week 24 | Baseline and week 24
  The DASS 21 is validated, self-reported scale. This scale comprises 21 questions using a 4-point Likert-type scale (0=not at all, 3=almost always), covering three dimensions mental health status. The total score of each dimension will be multiplied by two and scores ranged from 0 to 42.
Change from baseline in well-being on the KIDSCREEN-27 questionnaire at week 24 | Baseline and week 24
  The well-being will be measured by two domains of the KIDSCREEN-27 questionnaire, physical well-being consist 5-item and psychological with 7-item. For each item, participants respond using a scale with scores from one to five points.
Change from baseline in sleep on the Pittsburgh Sleep Quality Index (PSQI) at week 24 | Baseline and week 24
  The PSQI is a self-reported questionnaire that asks respondents to report on their sleep quality and signs of sleep disturbance for the 1-month period prior to completing the questionnaire. The PSQI includes 19 questions, categorized into seven groups (sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medications and daytime dysfunction). Each constituent question produces a score on a 4-point Likert-type scale (from 0 to 3) and the total score is made up of scores from each of the seven subgroups of questions, giving a cumulated score between 0 and 21.
Change from baseline in symptoms of mental health disorder on the Strengths and Difficulties Questionnaire' (SDQ) at week 24 | Baseline and week 24
  The SDQ The questionnaire has 25 items which comprise five domains, covering 2 subscales (ie, difficulties and strengths). The difficulties subscale consists of four domains: (i) emotional symptoms; (ii) conduct problems; (iii) hyperactivity/inattention; (iv) peer relationship problems; and the strengths subscale consists of one domain (v) pro-social behaviour. For each item, participants respond using a 3-point scale (ie, 'not true'=0, 'somewhat true'=1 and 'certainly true'=2) and each of the five subscales the score can range from 0 to 10. Lower scores indicate fewer psychological difficulties.
Process evaluation - consent rate | week 24
  The consent rate (% percentage) will be used to assess feasibility based on how many participants offered the program agreed to be involved. 2) retention rate (retention rate at 16 - wk follow-p); 3) attendance (student participation in the structured physical activity), 4) students´ satisfaction with the program ("I enjoyed participating in the RT sessions on 5-point Likert scale: 5=strongly agree to 1=strongly disagree) and 5) engagement ( student engagement with the pedometer self-monitoring and adherence to goals setting).
Process evaluation - retention rate | week 24
  The feasibility of the ActTeens Program will be assessed by retention rate (% percentage) at week 16; 3) attendance (student participation in the structured physical activity), 4) students´ satisfaction with the program ("I enjoyed participating in the RT sessions on 5-point Likert scale: 5=strongly agree to 1=strongly disagree) and 5) engagement ( student engagement with the pedometer self-monitoring and adherence to goals setting).
Process evaluation - Attendance | week 24
  The feasibility of the ActTeens Program will be assessed by attendance (% percentage) based on number of student participation in the structured physical activity. 4) students´ satisfaction with the program ("I enjoyed participating in the RT sessions on 5-point Likert scale: 5=strongly agree to 1=strongly disagree) and 5) engagement ( student engagement with the pedometer self-monitoring and adherence to goals setting).
Process evaluation - Satisfaction | week 24
  The students´ satisfaction (score) with the program will be assessed based on the following question :"I enjoyed participating in the RT sessions on 5-point Likert scale: 5=strongly agree to 1=strongly disagree.
Process evaluation - Engagement | week 24
  The student engagement with the pedometer self-monitoring (% percentage) and adherence to goals setting (% percentage) will be to assess feasibility of the ActTeens Program.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Stabelini Neto, PhD, Study Chair — Universidade Estadual do Norte do Parana; Géssika Castilho dos Santos, Ms, Principal Investigator — Universidade Estadual de Londrina
Locations (1):
- Universidade Estadual do Norte do Paraná, Jacarezinho, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The plan is to allow other researchers to use the data obtained in the study is this is approved byut the corresponding responsible persons.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: At the end of the trial.
Access Criteria: Approval of an analysis protocol by the study's steering committee

REFERENCES:
- [Derived] Stabelini Neto A, Santos GCD, Silva JMD, Correa RC, da Mata LBF, Barbosa RO, Zampier Ulbrich A, Kennedy SG, Lubans DR. Improving physical activity behaviors, physical fitness, cardiometabolic and mental health in adolescents - ActTeens Program: A protocol for a randomized controlled trial. PLoS One. 2022 Aug 9;17(8):e0272629. doi: 10.1371/journal.pone.0272629. eCollection 2022. PMID 35944003